CLINICAL TRIAL: NCT04956991
Title: Applications of CT in Differentiating Crohn's Disease Activity
Brief Title: CT Diagnoses in Crohn"s Disease Activity
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018130
Record Dates: First submitted 2021-06-29; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CDAI≤220: According to the Crohn's disease activity index (CDAI) scores, all the patients included in the study were divided into group A (CDAI≤220)
- CDAI>220: According to the Crohn's disease activity index (CDAI) scores, all the patients included in the study were divided into group B (CDAI>220)

SUMMARY:
The study focused on the clinical value of CT in assessing the activity of Crohn's disease.

DETAILED DESCRIPTION:
"Crohn's disease is an inflammatory disease with non-specific clinical manifestations. The lesions are more common in the ileocecal area and the end of the ileum, and also can affect the entire digestive tract. In recent years, the domestic incidence of Crohn's disease has been increasing. At present, CT diagnosis still lacks the gold standard and requirescombination of clinical manifestations, endoscopic examination, imaging examination and laboratory examination results. CT has showed advantages of non-invasive inspection, fast imaging speed, high tissue density resolution, and strong patient acceptability. In addition, the examination can clearly show the internal and external tissue structure of the digestive tract, which has been widely used in the diagnosis and activity evaluation of Crohn's disease.

In order to clarify the clinical value of CT in assessing the activity of Crohn's disease, this study mainly used retrospective analysis of the CT manifestations and clinical data of patients with Crohn's disease to explore the clinical value of CT in assessing the activity of patients with Crohn's disease."

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease patients with confirmed endoscopic or pathological examination results
* Complete laboratory data such as CRP, erythrocyte sedimentation rate, etc.

Exclusion Criteria:

* Related inspection results are not complete
* The interval between endoscopic and laboratory examination results exceeds 2 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Crohn"s disease with complete CT and clinical data
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Crohn's disease activity index (CDAI) scores | 1year
  Crohn's disease activity index (CDAI) scores

CONTACTS AND LOCATIONS:
Overall Officials: Jianyu Liu, Study Director — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No